CLINICAL TRIAL: NCT04252001
Title: Growing up With the Young Endocrine Support System (YESS!): Innovative E-technology to Improve Transition From Paediatric to Adult Care
Brief Title: Growing up With the Young Endocrine Support System (YESS!)
Acronym: YESS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: dr. Laura C. G. de Graaff-Herder (Other)
Responsible Party: Sponsor-Investigator, dr. Laura C. G. de Graaff-Herder, Principal Investigator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NL.69953.078.19; NL8097 (Other: Netherlands Trial Register)
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Congenital Adrenal Hyperplasia; Hypogonadotropic Hypogonadism; Growth Hormone Deficiency; Combined Pituitary Hormone Deficiency; Turner Syndrome; Klinefelter Syndrome; Addison's Disease; Androgen Insensitivity Syndrome; Thyroid Dysgenesis
Keywords: Serious game; Endocrinology; Transition
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Hypogonadism; Dwarfism, Pituitary; Combined Pituitary Hormone Deficiency; Turner Syndrome; Klinefelter Syndrome; Addison Disease; Androgen-Insensitivity Syndrome; Thyroid Dysgenesis

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group YT (Experimental): Group receives YESS! game and transition-toolkit
  Interventions: Device: YESS! game; Other: Transition-toolkit
- Group GT (Experimental): Group receives control game and transition-toolkit
  Interventions: Device: Snake '97; Other: Transition-toolkit
- Group T (Experimental): Group receives transition-toolkit
  Interventions: Other: Transition-toolkit
- Group O (No Intervention): Group receives usual transition care

INTERVENTIONS:
Device: YESS! game — The YESS! game is a real-life game for smartphone or tablet in which the player has to solve a mystery. The adolescent plays an active role in the course of the story. This results in an interactive experience. During the game, the adolescent is challenged with regard to self-management and responsible behaviour in general life, with parallels to medical selfmanagement and responsible behaviour.
  The adolescent has to decide at several different moments whether to take action or not, whether to accept help or not and whether to share (fictive) confidential information or not. Other aspects that are covered are 'taking responsibility' and 'being on time'. The choices the adolescent makes throughout the game are registered in a coded manner, for later analysis. The game is available in Dutch, English and Spanish.
  Arms: Group YT
Device: Snake '97 — Snake '97 is a game for smartphone or tablet which is free and can be downloaded in the App Store. The game is a remake of the original snake on the mobile phone in 1997 in which the player moves the snake around and makes the snake 'consume food' (little dots) which causes the snake to grow longer. The goal is to make the snake as large as possible. The game has 12 difficulty levels.
  Other Names: control game
  Arms: Group GT
Other: Transition-toolkit — The transition toolkit consists of paper cards with assignments, ideas and tips regarding medical self-management.
  Arms: Group GT; Group T; Group YT

SUMMARY:
Transition from paediatric to adult endocrinology is a challenge for adolescents, families and doctors. Up to 25% of young adults with chronic endocrine disorders are lost to follow-up ('drop-out') once the young adult moves out of paediatric care. Non-attendance and sub-optimal medical self-management can lead to serious and expensive medical complications. In a pilot study, adolescents suggested the use of e-technology to become more involved in the transition process. The investigators have designed and developed the YESS! game, a tool to help improve medical self-management in adolescents with chronic endocrine disorders. The hypothesis is that adolescents playing the YESS! game will show a larger increase in self-management score during the first year of transition and will have a lower drop-out rate at the adult endocrine outpatient clinic (OPC), compared to adolescents who do not play the game.

DETAILED DESCRIPTION:
Rationale: Transition from paediatric to adult endocrinology is a challenge for adolescents, families and doctors. Up to 25% of young adults with chronic endocrine disorders are lost to follow-up ('drop-out') once the young adult moves out of paediatric care. Non-attendance and sub-optimal medical self-management can lead to serious and expensive medical complications. In a pilot study, adolescents suggested the use of e-technology to become more involved in the transition process. The investigators have designed and developed the YESS! game, a tool to help improve medical self-management in adolescents with chronic endocrine disorders. The hypothesis is that adolescents playing the YESS! game will show a larger increase in self-management score during the first year of transition and will have a lower drop-out rate at the adult endocrine outpatient clinic (OPC), compared to adolescents who do not play the game.

Objective: 1.To improve medical self-management. 2.To prevent drop-out from the adult outpatient clinic. Study design: multicentre randomized controlled trial Study population: 160 transition patients from 15 to 20 years old from the participating countries Spain, The United Kingdom, Belgium and the Netherlands. Patients are diagnosed with a chronic endocrine disorder. Intervention: The study consists of 4 study arms: receiving the YESS! game and toolkit (group YT), receiving the control game and toolkit (group GT), receiving the toolkit only (group T) and receiving regular transition care (group O). Every group will receive regular transition care. The transition toolkit consists of paper cards with assignments, ideas and tips regarding medical self-management. Main study parameters: Primary outcome: the Self-management and Transition to Adulthood with Rx (=treatment) (STARx) questionnaire score 12 months after inclusion in group YT compared to group O. Secondary outcome: the STARx questionnaire score 6 months after inclusion in group YT compared to the other study groups, the STARx questionnaire score 12 months after inclusion in group YT compared to group GT and T and the drop-out rate to the adult outpatient clinic in the first year after the last visit to the paediatric endocrinologist (i.e. one year after the moment of transfer) in group YT compared to groups GT, T and O.

Nature and extent of the burden and risks associated with participation: The participants are not exposed to any risks. The YESS! and the control game are safe apps played on a mobile phone or tablet. The burden consists of filling out the STARx questionnaires and playing the YESS! or control game. The questionnaires will be filled out online at home at the start of the study and after 6 and 12 months. Every 6 months the subject has an appointment at the outpatient clinic. The participant can play the YESS! game for a maximum of 15 minutes a day to prevent game addiction. The control game could be played for an unlimited amount of time, but will unlikely cause game addiction since the game is not considered challenging and exciting enough.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 to 20 years old.
* Diagnosed with congenital adrenal hyperplasia, hypogonadotropic hypogonadism, Turner syndrome, Klinefelter syndrome, growth hormone deficiency, combined pituitary hormone deficiency, Androgen insensitivity syndrome, thyroid dysgenesis or Addison's disease

Exclusion Criteria:

* Lack of a mobile phone or tablet.
* Intellectual disability or language barrier leading to inability to use the YESS! game or the control game.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Medical self-management group YT compared to group O @12months | 12 months
  The difference in Self-management and Transition to Adulthood with Rx (treatment) (STARx) questionnaire score from baseline after 12 months in participants receiving the YESS! game and toolkit (group YT) compared to participants receiving regular care (group O).

SECONDARY OUTCOMES:
Medical self-management group YT compared to group GT and -T @12months | 12 months
  The difference in Self-management and Transition to Adulthood with Rx (treatment) (STARx) questionnaire score from baseline after 12 months in participants receiving the YESS! game and toolkit (group YT) compared to participants receiving the control game and toolkit (group GT) and participants receiving the toolkit only (group T).
  Transition to Adulthood with Rx (treatment) (STARx) questionnaire score in group YT compared to group GT and group T after 12 months.
Medical self-management in group YT compared to group GT, -T and -O @6months | 6 months
  The difference in Self-management and Transition to Adulthood with Rx (treatment) (STARx) questionnaire score from baseline after 6 months in participants receiving the YESS! game and toolkit (group YT) compared to participants receiving the control game and toolkit (group GT), participants receiving the toolkit only (group T) and participants receiving regular care (group O).
Drop-out rate adult outpatient clinic | 12 months
  The difference in the drop-out rate to the outpatient clinic in group YT compared to group GT, group T and group O during the first year after the last visit to the paediatric endocrinologist (i.e. one year after the moment of transfer, t=24 m).

CONTACTS AND LOCATIONS:
Overall Officials: Laura CG de Graaff, MD PhD, Principal Investigator — Erasmus Medical Centre
Locations (7):
- Ghent University Hospital, Ghent, Belgium
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands
- Hospital Infantil Universitario Niño Jesús, Madrid, Spain
- United Kingdom (4):
  - Queen Elizabeth University Hospital, Glasgow
  - Royal Hospital for Children, Glasgow
  - The Royal London Hospital (Barts Health NHS Trust), London
  - University College London Hospital (UCL Institute of Child Health), London

IPD SHARING:
Plan to Share IPD: Yes
The IPD has not been finalized yet. The investigators intent to share the full anonymized dataset, study protocol and statistical analysis plan upon request after publication of the results. Informed consent forms will not be shared."